CLINICAL TRIAL: NCT05198219
Title: Procedural Efficiency and Organisational Impact of Rhino Laryngoscopes Procedures in Consults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ambu A/S (Industry)
Collaborators: Sahlgrenska University Hospital (Other); Skane University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HE001
Record Dates: First submitted 2021-11-05; First posted 2022-01-20 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Laryngeal Disease
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rhinolaryngoscope Ambu® aScope™ 4 Rhinolaryngo (Experimental): All approved procedures performed during the study period.
  Interventions: Device: Ambu® aScope™ 4 Rhinolaryngo
- Conventional reusable rhinolaryngoscope (Active Comparator): All procedures performed during the study period.
  Interventions: Device: Conventional reusable rhinolaryngoscope

INTERVENTIONS:
Device: Ambu® aScope™ 4 Rhinolaryngo — Patient indication following a rhinolaryngoscopy
  Arms: Rhinolaryngoscope Ambu® aScope™ 4 Rhinolaryngo
Device: Conventional reusable rhinolaryngoscope — Patient indication following a rhinolaryngoscopy
  Arms: Conventional reusable rhinolaryngoscope

SUMMARY:
The aim of this study is to investigate the procedure efficiency, organisational and economic impact, and physician evaluation of the conventional reusable rhino laryngoscope vs. Ambu® aScope™ 4 RhinoLaryngo in procedures conducted distally form the ENT department e.g. in the emergency department (ED), intensive care unit (ICU), ward etc., i.e. consults.

DETAILED DESCRIPTION:
The aim of this study is to investigate the procedure efficiency, organisational and economic impact, and physician evaluation of the conventional reusable rhinolaryngoscope vs. Ambu® aScope™ 4 RhinoLaryngo in procedures conducted distally from the ENT department e.g. in the emergency department, intensive care unit, ward etc., i.e. consults.

The study will be prospective and randomised until 13 procedures have been performed in each group followed by an assessment of the organisational impact and cost comparison of the two technologies. The investigator will track the time and evaluate the device after each procedure. The organisational impact will be accessed by a questionnaire following the study period. A cost comparison will be enabled via tracking all the processes associated with the rhinolaryngoscopes. After tracking all equipment, time, and utilities will be ascribed a cost.

ELIGIBILITY:
Inclusion Criteria:

* The investigator has been trained and conducted at least 5 successful training procedures with both the aScope 4 RhinoLaryngo and the reusable rhinolaryngoscope systems.
* The investigator on call for consults must be available to fill out the CRF immediately before and after the procedure.
* The investigator must be dedicated to the study while on call for consults
* Clinical indication and eligible for a rhino laryngoscopy, as judged by the physician
* Patients ≥18 years

Exclusion Criteria:

* If the patient has no clear indication for rhino laryngoscopy the procedure should not be conducted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Pre-procedure time from notification of the physician to start of rhinolaryngoscopy. | Prior to procedure
  The time (minutes) from indication of the need for a rhinolaryngoscopy, as registered by the physician until initiation of rhinolaryngoscopy. The mean time registered for the experimental arm will be compared to the active comparator arm to assess differences.

SECONDARY OUTCOMES:
Availability assessed as the time from indication of the need of the rhinolaryngoscopy until the physician leaves to conduct the rhinolaryngoscopy. | Prior to procedure
  Time (minutes) from indication of the need for rhinolaryngoscopy until the investigator leave to conduct the rhinolaryngoscopy. The mean time registered for the experimental arm will be compared to the mean time registered for the active comparator arm to assess differences.
Time from indication for the need of rhinolaryngoscopy until the procedure is completed. | Within 24 hours after completion of procedure.
  Time from indication for the need of rhinolaryngoscopy until the rhinolaryngoscope has been fully removed from the patient.
  The outcome will be reported as the area under the curve compared between experimental and active comparator arm.
Organisational impact - User preference for type of rhinolaryngoscope assessment of work process. | Up to 26 weeks after study completion
  User preference assessment of parameters for rhinolaryngoscopy work process (1. Free of wear and tear, 2. Training and education of students, 3. Recording and saving images and videos). Responses rated through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope for workflow. | Up to 26 weeks after study completion
  Comparison between workflows for the experimental arm or active comparator. Assessed as the preference of the treating physician through a 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User evaluation for type of rhinolaryngoscope based on time until start of rhinolaryngoscopy. | Up to 26 weeks after study completion
  User evaluation of which rhinolaryngoscope is expected to have the longest time interval from indication for rhinolaryngoscopy until the start of the procedure, based on previous experience.
  Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope based on patient/carer involvement in procedure. | Up to 26 weeks after study completion
  User assessment of which rhinolaryngoscope is the most cumbersome to involve patients or carers in the procedure and subsequent diagnosis or clinical decision (e.g. show or present the procedure and findings during or following the procedure).
  Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact- User preference for type of rhinolaryngoscope based on training requirements and skills. | Up to 26 weeks after study completion
  User preference of training requirement and skills needed from health-care professionals to maneuver rhinolaryngoscope.
  Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope based on modes of operation | Up to 26 weeks after study completion
  User preference of which rhinolaryngoscope requires most coordination with colleagues to ensure ready-to-use rhinolaryngoscopes.
  Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope based on vigilance and monitoring methods. | Up to 26 weeks after study completion
  User preference of which rhinolaryngoscope requires the least vigilance and monitoring of high hazard or highly infectious diseases.
  Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope based on working conditions and safety. | Up to 26 weeks after study completion
  User preference of which rhinolaryngoscope makes the user feel most exposed to infectious agents. Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - Hospital management preference for type of rhinolaryngoscope based on budget allocation. | Up to 26 weeks after study completion
  Hospital management preference for which rhinolaryngoscope requires the least complex budgeting to ensure patient-ready endoscopes and associated technologies. Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Organisational impact - User preference for type of rhinolaryngoscope based on logistics. | Up to 26 weeks after study completion
  User preference of which rhinolaryngoscope is associated with the biggest logistical burden. Response through 3-point scale - favorable to: 1. Ambu single-use rhinolaryngoscope or 2. conventional reusable rhinolaryngoscope or 3. neutral. Results distributed in percentages.
Perception of device | During procedure
  User preference of the image quality, maneuverability, ergonomics of the handle and overall perception of quality of the rhinolaryngoscope will be assessed through a 5-point Likert scale (very poor, poor, acceptable, good or very good).
Intended device | During procedure
  Conversion rate from the rhinolaryngoscope initially intended for the procedure to another rhinolaryngoscope.
Rate of complications | During procedure
  Rate of complications or issues with the rhinolaryngoscope or associated technologies.
Frequency of procedures | Assessed no more than 48 hours after completed week.
  Total number of procedures performed per week compared between experimental arm and active comparator.

CONTACTS AND LOCATIONS:
Overall Officials: Johan Hellgren, MD, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Ambu A/S, Ballerup Municipality, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gudnadottir G, Hafsten L, Dahl Travis H, Nielsen K, Hellgren J. Comparison of utility and organizational impact of reusable and single-use rhinolaryngoscopes in a tertiary otorhinolaryngology department. Front Surg. 2024 Oct 7;11:1380571. doi: 10.3389/fsurg.2024.1380571. eCollection 2024. PMID 39435392